CLINICAL TRIAL: NCT00710788
Title: Interventional, Multicenter, Prospective, Randomized Trial to Slow Down the Progression of Cardiovascular Calcifications to Reduce QTd in Incident Dialysis Patients
Brief Title: Reduce Cardiovascular Calcifications to Reduce QT Interval in Dialysis
Acronym: Independent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria ASL Avellino 2 (Other)
Responsible Party: Principal Investigator, Dr Biagio Di Iorio, MD, PhD, Azienda Sanitaria ASL Avellino 2
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008.1; 2008.1.brd.renagel
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Cardiovascular Mortality
Keywords: QT interval; QT dispersion; arrhythmias; death; TC score
MeSH Terms: conditions — Arrhythmias, Cardiac; Death | interventions — Sevelamer; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): sevelamer as Phosphate-binder treatment
  Interventions: Drug: sevelamer phosphate-binders
- 2 (Active Comparator): Calcium carbonate
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: sevelamer phosphate-binders — 1600 mg/day for 2 years
  Other Names: Renagel
  Arms: 1
Drug: Calcium Carbonate — Calcium carbonate 1 g/day for 2 years
  Arms: 2

SUMMARY:
Research proposal to evaluate the impact of different phosphate binders on the progression of cardiovascular calcification and QT dispersion in new haemodialysis patients.

DETAILED DESCRIPTION:
The risk of developing cardiovascular diseases in patients on hemodialysis is higher than in general population. Higher levels of serum phosphate are associated with adverse cardiovascular outcomes, especially in the setting of overt hyperphosphatemia. Given the biological importance of serum phosphorus, it is conceivable that also within the normal range values the higher serum phosphate levels may be associated with the worst outcome. Several paper have shown that vascular calcifications in dialysis patients are associated with increased relative risk of death; it has also been demonstrated in uremic patients that vascular calcifications decrease arterial elasticity. We previously observed that vascular calcification directly correlate with QT interval (QTc) as well as QT dispersion (QTd) in dialysis. Also, QT correction (obtained by the correction of phosphoremia and dyslipidemia) can ameliorate the development of arrhythmia and sudden death. Aim of this study is to evaluate the relationship between vascular calcifications and both QTd increase and mortality in incident hemodialysis patients, and to investigate the efficacy of sevelamer to reduce vascular calcifications and QTd.

ELIGIBILITY:
Inclusion Criteria:

* incident patients on haemodialysis (CKD stage 5);
* an informed consent will be provided at the study entry.

Exclusion Criteria:

* congenital prolongation of QT segment syndrome;
* QTc >440 ms; increased QTd;
* bradycardia <50 bpm;
* sintomatic arrhythmia or any other significant heart problems;
* electrolyte unbalances (especially hypokalemia, hypomagnesemia, hypocalcemia);
* abnormal liver function tests;
* hypothyroidism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2007-01; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
death due to cardiac arrhythmias or as sudden cardiac death defined as any deaths coded as "cardiac arrest, cause unknown" or "cardiac arrhythmia" without any exclusions | 2 years

SECONDARY OUTCOMES:
QT interval; PWV; mortality for acute myocardial infarction, cerebral vascular accident and heart failure; Non-CV mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Biagio R Di Iorio, MD, PhD, Study Chair — ASL AV/2, Avellino, Italy; Loreto Gesualdo, professor, Principal Investigator — Nephrology Division, Medical School, University of Foggia; Filippo Aucella, MD, Principal Investigator — ASL FG, Italy; Walter De Simone, MD, Principal Investigator — AO MOscati, Avellino, Italy; Mario Migliorati, MD, Principal Investigator — Dialysis, Torre del Greco, Italy; Domenico Santoro, MD, Principal Investigator — Nephrology Division, Medical School, University of Messina, Italy; Pasquale Guastaferro, MD, Principal Investigator — Nephrology Division, ASL AV1, Sant'Angelo de Lomnardi, Italy; Luigi Chiuchuilo, MD, Principal Investigator — Dialysis, Avellino, Italy; Vincenzo Tedesco, MD, Principal Investigator — Dialysis, Montella, Italy
Locations (1):
- Nephrology Division, Solofra, Avellino, Italy

REFERENCES:
- [Background] Di Iorio B, D'Avanzo E, Piscopo C, Cucciniello E, Bellizzi V: QT and phosphatemia: a novel sensitive marker of cardiovascolar risk for an old killer . 12th Assisi European Meeting on Cardionephrology, Cardionephrology 10, Nuova BIOS ed, 2008;23-26
- [Result] Marangon N, Lindholm B, Stenvinkel P. Nonphosphate-binding effects of sevelamer--are they of clinical relevance? Semin Dial. 2008 Sep-Oct;21(5):385-9. doi: 10.1111/j.1525-139X.2008.00440.x. Epub 2008 Jun 19. PMID 18573137
- [Result] Di Iorio BR, Bortone S, Piscopo C, Grimaldi P, Cucciniello E, D'Avanzo E, Mondillo F, Cillo N, Bellizzi V. Cardiac vascular calcification and QT interval in ESRD patients: is there a link? Blood Purif. 2006;24(5-6):451-9. doi: 10.1159/000095362. Epub 2006 Aug 25. PMID 16940716
- [Result] Di Iorio BR, D'Avanzo E, Piscopo C, Grimaldi P, Cucciniello E, Cillo N, Bellizzi V. Progression of vascular calcification increases QT interval in haemodialysis patients. Nephrol Dial Transplant. 2006 Dec;21(12):3609-10. doi: 10.1093/ndt/gfl417. Epub 2006 Jul 31. No abstract available. PMID 16880182
- [Result] Cozzolino M, Galassi A, Pasho S, Fallabrino G, Gallieni M, Brancaccio D. Preventive measures and new pharmacological approaches of calcium and phosphate disorders. Contrib Nephrol. 2008;161:234-239. doi: 10.1159/000130696. PMID 18451682
- [Result] Nolan CR, McCarron DA. Lack of mortality benefit with sevelamer. Kidney Int. 2008 May;73(9):1093; author reply 1093-4. doi: 10.1038/ki.2008.46. No abstract available. PMID 18414441
- [Result] Wrong O, Harland C. Sevelamer. Nephrol Dial Transplant. 2008 Jun;23(6):2108; author reply 2101-2. doi: 10.1093/ndt/gfn162. Epub 2008 Apr 9. No abstract available. PMID 18400812
- [Result] Negri AL. [K-DOQI guidelines for calcium and phosphorus metabolism in chronic kidney disease: outcomes, compliance and new drugs for treatment]. Nefrologia. 2007;27(6):670-3. No abstract available. Spanish. PMID 18336094
- [Result] Hamida FB, Fatma LB, Barbouch S, Kaaroud H, Helal I, Hedri H, Abdallah TB, Maiz HB, Kheder A. Effect of sevelamer on mineral and lipid abnormalities in hemodialysis patients. Saudi J Kidney Dis Transpl. 2008 Mar;19(2):183-8. PMID 18310864
- [Result] St Peter WL, Liu J, Weinhandl E, Fan Q. A comparison of sevelamer and calcium-based phosphate binders on mortality, hospitalization, and morbidity in hemodialysis: a secondary analysis of the Dialysis Clinical Outcomes Revisited (DCOR) randomized trial using claims data. Am J Kidney Dis. 2008 Mar;51(3):445-54. doi: 10.1053/j.ajkd.2007.12.002. PMID 18295060
- [Result] Winkelmayer WC, Tonelli M. Phosphate binder choice in dialysis patients: a call for evidence-based rather than marketing-based clinical practice. Am J Kidney Dis. 2008 Mar;51(3):362-5. doi: 10.1053/j.ajkd.2008.01.004. No abstract available. PMID 18295050
- [Result] Mansour J, Shahapuni I, El Esper N, Fournier A. Block randomized trial evidencing lower mortality with sevelamer compared with calcium phosphate binder in incident dialysis patients. Kidney Int. 2008 Feb;73(4):510. doi: 10.1038/sj.ki.5002752. No abstract available. PMID 18235525
- [Result] Ferreira A, Frazao JM, Monier-Faugere MC, Gil C, Galvao J, Oliveira C, Baldaia J, Rodrigues I, Santos C, Ribeiro S, Hoenger RM, Duggal A, Malluche HH; Sevelamer Study Group. Effects of sevelamer hydrochloride and calcium carbonate on renal osteodystrophy in hemodialysis patients. J Am Soc Nephrol. 2008 Feb;19(2):405-12. doi: 10.1681/ASN.2006101089. Epub 2008 Jan 16. PMID 18199805
- [Result] Suki WN; Dialysis Clinical Outcomes Revisited Investigators. Effects of sevelamer and calcium-based phosphate binders on mortality in hemodialysis patients: results of a randomized clinical trial. J Ren Nutr. 2008 Jan;18(1):91-8. doi: 10.1053/j.jrn.2007.10.019. PMID 18089452
- [Result] Russo D, Miranda I, Ruocco C, Battaglia Y, Buonanno E, Manzi S, Russo L, Scafarto A, Andreucci VE. The progression of coronary artery calcification in predialysis patients on calcium carbonate or sevelamer. Kidney Int. 2007 Nov;72(10):1255-61. doi: 10.1038/sj.ki.5002518. Epub 2007 Sep 5. PMID 17805238
- [Result] Suki WN, Zabaneh R, Cangiano JL, Reed J, Fischer D, Garrett L, Ling BN, Chasan-Taber S, Dillon MA, Blair AT, Burke SK. Effects of sevelamer and calcium-based phosphate binders on mortality in hemodialysis patients. Kidney Int. 2007 Nov;72(9):1130-7. doi: 10.1038/sj.ki.5002466. Epub 2007 Aug 29. PMID 17728707
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Ruggeri M, Bellasi A, Cipriani F, Molony D, Bell C, Russo D, Di Iorio B. Sevelamer is cost effective versus calcium carbonate for the first-line treatment of hyperphosphatemia in new patients to hemodialysis: a patient-level economic evaluation of the INDEPENDENT-HD study. J Nephrol. 2015 Oct;28(5):593-602. doi: 10.1007/s40620-014-0122-8. Epub 2014 Jul 16. PMID 25027030
- [Derived] Di Iorio BR, Cucciniello E, Bellizzi V. Vascular calcification and QT interval in incident hemodialysis patients. J Nephrol. 2009 Nov-Dec;22(6):694-8. PMID 19967647